CLINICAL TRIAL: NCT00526877
Title: Evaluation of Efficacy and Safety of Long-acting Risperidone Microspheres in Patients With Schizophrenia or Schizoaffective Disorders, Who is Receiving Psychiatric Home-care Treatment, When Switching From Typical Depot or Oral Antipsychotics to Long-acting Risperidone Microspheres
Brief Title: An Efficacy and Safety Study of Long-acting Risperidone in Participants With Schizophrenia or Schizoaffective Disorders Who Are Receiving Psychiatric Home Care Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013873; RISSCH4119
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Schizophrenia; Schizoaffective Disorders
Keywords: Schizophrenia; Schizoaffective disorders; Risperidone; Risperdal Consta
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Risperidone (Experimental): Risperidone long-acting injectable 25 milligram (mg) or 37.5 mg or 50 mg will be administered intramuscularly (into a muscle) depending on Investigator's discretion every 2 weeks for 24 weeks.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Risperidone — Risperidone long-acting injectable 25 milligram (mg) or 37.5 mg or 50 mg will be administered intramuscularly (into a muscle) depending on Investigator's discretion every 2 weeks for 24 weeks.
  Other Names: Risperdal Consta

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of long-acting risperidone microspheres (small uniformly-sized spherical particles, of micrometer dimensions, frequently labeled with radioisotopes or various reagents acting as tags or markers) in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self) and schizoaffective disorders (a mixed psychiatric disorder relating to a complex psychotic state that has features of both schizophrenia and a mood disorder such as bipolar disorder), who are receiving psychiatric home-care treatment .

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-centric (conducted in more than one center), non-randomized and single-arm study of long- acting risperidone microspheres in participants with schizophrenia and schizoaffective disorders. The duration of this study will be 6 months and will include following parts: Screening (that is, 28 days before study commences on Day 1), run-in period (that is, Week 1 to 3) and Treatment period (that is, Week 1 to 24). Participants will receive previous medication for the first three weeks during run-in period and previous medications will be tapered off during the third week. Participants will receive long-acting risperidone microspheres starting at a dose of 25 milligram (mg) every two weeks by intramuscular injection (injection of a substance into a muscle). Efficacy of the participants will be primarily evaluated through Positive and Negative Syndrome Scale.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for schizophrenia or schizoaffective disorder according to Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV)
* Participant has been given an adequate dose of an appropriate antipsychotic for an adequate period of time prior to enrollment, but previous treatment is considered unsatisfactory due to one or more of the following reasons: lack of efficacy, lack of tolerability or safety, lack of compliance and/or other reasons to switch to another antipsychotic medication
* Female participants must be postmenopausal, surgically sterile, or practicing an effective method of birth control before entry and throughout the study; have a negative urine betahuman chorionic gonadotropin (HCG) pregnancy test at screening; and a negative urine pregnancy test on screening visit
* Participants or their legally acceptable representatives must have signed an informed consent document

Exclusion Criteria:

* Participants with a primary, active DSM-IV diagnosis other than schizophrenia and schizoaffective disorder
* Participants with relevant history or current presence of any significant and/or unstable cardiovascular, respiratory, neurological (including seizures or significant cerebrovascular), renal, hepatic, hematologic, endocrine, immunologic or other systemic disease
* Participants that are previously on concomitant use of Risperdal CONSTA
* History or current symptoms of tardive dyskinesia
* History of neuroleptic malignant syndrome (NMS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Positive and Negative Syndromes Scale (PANSS) Total Score at Week 24 | Baseline and Week 24
  The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening.

SECONDARY OUTCOMES:
Personal and Social Performance (PSP) Scale Score | Screening (28 days before study drug administration), Baseline and Week 24
  The PSP is a clinician-rated scale that reflects social functioning in 4 domains of behavior (socially useful activities including work and study, personal and social relationships, self care, and disturbing and aggressive behaviors). The total score ranges from 1 to 100 (score of 71 to 100 will have a mild degree of difficulty; from 31 to 70, varying degrees of disability; less than or equal to 30, functioning so poorly as to require intensive supervision) divided into 10 equal intervals to rate the degree of difficulty (i=absent to vi=very severe) in each of the 4 domains.
Clinical Global Impression (CGI) Scale Score | Screening (28 days before study drug administration), Baseline and Week 24
  The CGI rating scale is a 7-point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 indicates to "normal, not at all ill" and a rating of 7 indicates "among the most extremely ill participants". Higher scores indicate worsening.
Short Form-36 (SF-36) - Quality of Life Score | Screening (28 days before study drug administration), Baseline and Week 24
  The SF-36 is a survey of participant health. It consists of eight scaled scores, which are the weighted sums of the questions in their section. The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Each item is scored on a 0-100 range so that the lowest and highest possible scores are set at 0 and 100, respectively. All items are scored so that a high score defines a more favorable health state.
Change From Baseline in Simpson Angus Rating Scale (SAS) Score at Week 24 | Baseline and Week 24
  The SAS rates 10 items from 0 (normal) to 4 (extreme), including gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, leg pendulousness, head rotation, Glabellar tap, tremor and salivation. The SAS global score is the average score (total sum of items score divided by the number of items) and ranges between 0 and 4, where the higher score denotes more severe condition of extra pyramidal symptoms.
Change From Baseline in Extrapyramidal Symptoms Rating Scale (ESRS) Total Score at Week 24 | Baseline and Week 24
  The ESRS is used to assess four types of drug-induced movement disorders administered as a questionnaire. Score range from 0 to 6 (0 is absent and 6 is extremely severe).
Number of Participants Compliant With Study Treatment | 6 months before administration of study drug and 6 months after administration of study drug
  Participants compliant with study treatment will be the participants who will complete the study treatment regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan, Ltd. Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd

REFERENCES:
- See also: An Efficacy and Safety Study of Long-acting Risperidone in Participants with Schizophrenia or Schizoaffective disorders who are Receiving Psychiatric Home Care Treatment — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=696&filename=CR013873_CSR.pdf